CLINICAL TRIAL: NCT01159743
Title: A Comparison of Body Fat Distribution in HIV-1 Infected Patients Receiving, Since the Beginning and for at Least Two Years, an Antiretroviral Therapy Based on Efavirenz or Lopinavir/Ritonavir Combined With Tenofovir + Emtricitabine or Lamivudine
Acronym: LYNX
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Demométrica (Unknown)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-031
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: HIV Infection
Keywords: lipodystrophy; Lipoatrophy; antiretroviral treatment
MeSH Terms: conditions — HIV Infections; Lipodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Efavirenz: HIV-infected patients on initial antiretroviral therapy for at least two years with efavirenz (Sustiva®; EFV) with a combination of tenofovir (TDF) plus emtricitabine (FTC) or lamivudine (3TC).
- Lopinavir / Ritonavir: HIV-infected patients on initial antiretroviral therapy for at least two years with lopinavir/ritonavir (Kaletra®; LPV/r) with a combination of tenofovir (TDF) plus emtricitabine (FTC) or lamivudine (3TC).

SUMMARY:
The purpose of this study is to compare the body fat distribution in Human Immunodeficiency Virus-1 (HIV-1) infected patients receiving, since the beginning and for at least two years, an antiretroviral therapy based on efavirenz or lopinavir/ritonavir and a combination of tenofovir plus emtricitabine (or lamivudine).

DETAILED DESCRIPTION:
Lipodystrophy (also called abnormal fat redistribution) associated with HIV infection is characterized by loss of subcutaneous adipose tissue (lipoatrophy) that is more apparent in the limbs, face, and buttocks, or by accumulation of adipose tissue (lipohypertrophy) in the intra-abdominal cavity, the mid, upper back, and breasts. Lipodystrophy may also occur in a mixed form (lipoatrophy and lipohypertrophy in the same patient).

Participants made a single study visit. Dual energy X-ray absorptiometry (DEXA) was performed within 30 days of this study visit. In addition, routine visit clinical results, demographic data, disease data, comorbidities and concomitant medications were collected.

ELIGIBILITY:
Inclusion Criteria

* Men and women aged ≥ 18 years with HIV-1 infection who are clinically stable and who were invited to participate in the study at a routine follow-up visit.
* HIV-1 infected patients receiving since the beginning and continuously, for at least two years, initial antiretroviral therapy (ART) based on efavirenz (EFV) and a combination of tenofovir (TDF) + emtricitabine (FTC) [or lamivudine (3TC)] or HIV-1 infected patients receiving since the beginning and continuously, for at least two years, initial ART based on lopinavir/ritonavir (LPV/r) and a combination of TDF +FTC (or 3TC).
* Patients with an undetectable viral load, in response to the detection limit of each participating hospital defined in the last 6 months.
* Patients who have given written informed consent to participate in this study [personal data collection and performance of dual energy X-ray absorptiometry (DEXA)].

Exclusion Criteria

* Patients who have received at some point both efavirenz (EFV) and lopinavir/ritonavir (LPV/r) in combination regimen or thereafter.
* Patients who have had structured treatment interruptions (therapeutic holidays).
* Patients with a body mass index <16 kg/m^2.
* Patients with metallic prostheses or prosthetic material that could interfere with the measurement of dual energy X-ray absorptiometry (DEXA).
* Patients with a history of plastic or repair surgery in the buttocks and breasts.
* Patients with a diagnostic test with barium or radionucleotides, performed during the last month.
* Pregnant women.
* Patients treated with other agents under investigational phase.
* Patients on current treatment with systemic corticosteroids or chemotherapy.
* Diabetes mellitus and hypoglycaemic treatment.
* Transsexualism (though implicit in prostheses and drugs).
* Any drug taken chronically, which may alter the distribution of fat or adipocyte biology (insulin, non-steroidal anti-inflammatory drugs, etc).
* Patient has undergone liposuction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients visiting Spanish HIV clinics.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Burgos, Other, Study Director — Abbvie Farmaceutica S.L.U. Spain
Locations (26):
- Spain (26):
  - Site Reference ID/Investigator# 39595, Alicante
  - Site Reference ID/Investigator# 39602, Barcelona
  - Site Reference ID/Investigator# 39605, Barcelona
  - Site Reference ID/Investigator# 39589, Barcelona
  - Site Reference ID/Investigator# 39601, Barcelona
  - Site Reference ID/Investigator# 39593, Barcelona
  - Site Reference ID/Investigator# 39603, Barcelona
  - Site Reference ID/Investigator# 39587, Bilbao
  - Site Reference ID/Investigator# 39596, Cabuenes-Gijon
  - Site Reference ID/Investigator# 39592, Donostia / San Sebastian
  - Site Reference ID/Investigator# 39590, Granada
  - Site Reference ID/Investigator# 39604, La Laguna Teneriffe
  - Site Reference ID/Investigator# 39609, Logroño
  - Site Reference ID/Investigator# 39597, Madrid
  - Site Reference ID/Investigator# 39600, Madrid
  - Site Reference ID/Investigator# 39591, Madrid
  - Site Reference ID/Investigator# 24822, Madrid
  - Site Reference ID/Investigator# 39586, Madrid
  - Site Reference ID/Investigator# 39599, Madrid
  - Site Reference ID/Investigator# 39611, Madrid
  - Site Reference ID/Investigator# 39588, Málaga
  - Site Reference ID/Investigator# 39606, Seville
  - Site Reference ID/Investigator# 39598, Valencia
  - Site Reference ID/Investigator# 39612, Valencia
  - Site Reference ID/Investigator# 39607, Vigo
  - Site Reference ID/Investigator# 39610, Zaragoza

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Efavirenz: Human Immunodeficiency Virus 1 (HIV-1)-infected patients on initial and continuous antiretroviral therapy for at least two years with efavirenz (Sustiva®; EFV) with a combination of tenofovir (TDF) plus emtricitabine (FTC) or lamivudine (3TC).
- Lopinavir / Ritonavir: HIV-infected patients on initial and continuous antiretroviral therapy for at least two years with lopinavir/ritonavir (Kaletra®; LPV/r) with a combination of tenofovir (TDF) plus emtricitabine (FTC) or lamivudine (3TC).
Period: Overall Study
Arm/Group | Efavirenz | Lopinavir / Ritonavir
Started | 237 | 109
Completed | 237 | 109
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efavirenz | Lopinavir / Ritonavir | Total
Number analyzed (Participants) | 237 | 109 | 346
Age Continuous [Mean (Standard Deviation); unit: years] — Data available for 235 and 109 patients in each treatment group respectively, 344 total patients.
  years | 42.2 (9.74) | 44.3 (9.46) | 42.8 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 17 | 55
  Male | 199 | 92 | 291
Region of Enrollment [Number; unit: participants]
  Spain | 237 | 109 | 346
Hepatitis C Virus (HCV) Co-infection [Number; unit: participants]
  HCV positive | 41 | 33 | 74
  HCV negative | 196 | 76 | 272
Time on current antiretroviral regimen [Number; unit: participants]
  2 - 3 years | 75 | 27 | 102
  3 - 4 years | 76 | 32 | 108
  More than 4 years | 86 | 50 | 136
Undetectable HIV-1 RNA (< 50 copies/mL) [Number; unit: participants] — Data available for 236 and 109 patients in each treatment group respectively, 345 total patients.
  participants | 236 | 109 | 345
Cluster of differentiation 4 (CD4)+ T-cell count [Mean (Standard Deviation); unit: cells/µL] — Data available for 236 and 108 patients in each treatment group respectively, 344 total patients.
  cells/µL | 585.56 (246.87) | 592.75 (258.77) | 587.82 (250.31)
CD4+ T-cell count nadir [Mean (Standard Deviation); unit: cells/µL] — Data available for 231 and 107 patients in each treatment group respectively, 338 total patients.
  cells/µL | 216.85 (121.88) | 169.94 (153.84) | 202.00 (134.39)
Previous acquired immunodeficiency syndrome (AIDS) diagnosis [Number; unit: participants] — Data available for 237 and 108 patients in each treatment group respectively, 345 total patients.
  participants
    Yes | 39 | 34 | 73
    No | 198 | 74 | 272

OUTCOME MEASURES:

1. Primary Outcome: Total Limb Fat Mass
Description: Total limb fat mass was assessed by dual energy X-ray absorptiometry (DEXA) scan. DEXA uses a whole body scanner and two different low-dose x-rays to read bone mass and soft tissue mass.
Time Frame: Study visit
Population: All participants for whom data were available.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Efavirenz | Lopinavir / Ritonavir
Number analyzed (Participants) | 232 | 106
kg | 8.84 (4.45) | 9.13 (6.26)

2. Secondary Outcome: Distribution of Body Fat Mass
Description: Body fat mass was assessed by dual energy X-ray absorptiometry (DEXA) scan.
Time Frame: Study visit
Population: All participants for whom data were available. The number of participants included in the analysis of each category for each group of participants is shown as "N" (EFV and then LPV/r).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Efavirenz | Lopinavir / Ritonavir
Number analyzed (Participants) | 237 | 109
kg
  Total body fat mass [N=231, 106] | 20.13 (7.56) | 20.24 (8.60)
  Trunk fat mass [N=232, 106] | 10.77 (4.84) | 10.76 (5.24)
  Upper limb fat mass [N=232, 106] | 2.11 (1.07) | 2.08 (1.14)
  Lower limb fat mass [N=232, 106] | 6.72 (3.68) | 7.04 (5.72)

3. Secondary Outcome: Lipodystrophy Severity Grading Scale (LSGS) Scores
Description: Perception of body fat was assessed by the Lipodystrophy Severity Grading Scale (LSGS), a standardized measurement of subjective lipoatrophy (fat loss) and lipoaccumulation (fat gain) perceived by the participant and by the physician. The degree of lipoatrophy and diffuse fat accumulation at each region was rated by both the participant and the physician as: Score 0=absent; Score 1=mild or noticeable on close inspection; Score 2=moderate or readily noticeable by patient/physician; Score 3=severe or readily noticeable to a casual observer.
  Score A reflects the lipoatrophy or fat loss perception at the face, arms, buttocks and legs and ranges from 0-12.
  Score B reflects the perception of fat gain at the abdomen, neck, and breasts and ranges from 0-9.
  The overall score is the sum of the scores A+B, and ranges from 0-21.
  Higher numbers indicate more fat loss (Score A) or gain (Score B). An average overall patient/physician score >7 indicates a clinical diagnosis of lipodystrophy.
Time Frame: Study visit
Population: All participants for whom data were available. The number of participants included in the analysis of each score for each group of participants is shown as "N" (EFV and then LPV/r).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Efavirenz | Lopinavir / Ritonavir
Number analyzed (Participants) | 237 | 109
units on a scale
  Patient Score A (fat loss) [N=233, 105] | 1.02 (1.92) | 1.12 (2.00)
  Patient Score B (fat gain) [N=235, 103] | 0.98 (1.50) | 1.17 (1.86)
  Patient Overall Score [N=233, 102] | 2.01 (2.68) | 2.33 (3.00)
  Physician Score A (fat loss) [N=233, 105] | 0.70 (1.27) | 1.04 (1.76)
  Physician Score B (fat gain) [N=235, 103] | 0.60 (1.10) | 0.76 (1.35)
  Physician Overall Score [N=233, 102] | 1.31 (1.80) | 1.83 (2.43)

4. Secondary Outcome: Change Over Time in Body Fat Distribution
Description: Change over time in total body fat and fat in the limbs and trunk was assessed by dual X-ray absorptiometry (DEXA) in participants for whom a DEXA measurement performed at least 6 months before participation in this study was available.
  A negative change score indicates fat loss over time and a positive change score indicates fat gain over time.
Time Frame: DEXA performed at the study visit and more than 6 months prior to the study visit (the period of time between the DEXA recorded at the study visit and the previous DEXA ranged from 6 to 36 months).
Population: Participants for whom a dual X-ray absorptiometry measurement performed at least 6 months before participation in this study was available.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Efavirenz | Lopinavir / Ritonavir
Number analyzed (Participants) | 34 | 14
kg
  Total fat mass | -0.05 (4.02) | -0.06 (7.34)
  Trunk fat mass | 0.32 (2.23) | -0.05 (4.04)
  Limb fat mass | 0.16 (2.43) | 0.10 (3.37)
  Upper limb fat mass | 0.39 (0.69) | -0.03 (0.66)
  Lower limb fat mass | 0.12 (2.13) | 0.13 (2.80)

ADVERSE EVENTS:
Arm/Group | Efavirenz | Lopinavir / Ritonavir
Serious Adverse Events (participants affected / at risk) | 0/237 | 0/109
Other Adverse Events (participants affected / at risk) | 0/237 | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.